CLINICAL TRIAL: NCT01509950
Title: Comparison of Staples Versus Nonabsorbable Subcuticular (Prolene) Suture for Skin Closure in Cesarean Deliveries: A Randomized Study
Brief Title: Comparison of Staples Versus Prolene Suture for Skin Closure at Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Natali Aziz, Clinical Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22389
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2018-11

CONDITIONS: Pregnancy; Cesarean Section
MeSH Terms: interventions — Sutures; glycolide E-caprolactone copolymer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Staples (Active Comparator): Use of staples for skin closure at cesarean section
  Interventions: Procedure: Staples
- Prolene non-absorbable sutures (Active Comparator): Use of Prolene non-absorbable sutures for skin closure at cesarean section
  Interventions: Procedure: Prolene non-absorbable sutures
- Absorbable sutures (Active Comparator): Use of absorbable sutures for skin closure at cesarean section; monocryl or vicryl.
  Interventions: Procedure: Absorbable Sutures

INTERVENTIONS:
Procedure: Staples — Staples for closure of cesarean section skin incision
  Other Names: Reflex one skin stapler 35 wide. Manufactured by Conmed
  Arms: Staples
Procedure: Prolene non-absorbable sutures — Prolene non-absorbable sutures for closure of cesarean skin incision
  Other Names: Prolene 2-0 18 inch on FS needle. Manufactured by Ethicon
  Arms: Prolene non-absorbable sutures
Procedure: Absorbable Sutures — Absorbable sutures for closure of cesarean skin incision
  Other Names: Monocryl or Vicryl. Manufactured by Ethicon
  Arms: Absorbable sutures

SUMMARY:
Currently different materials are used to close the skin after a cesarean delivery, including absorbable suture, non-absorbable suture and staples. It is not known what is the best choice of material to close the skin after a cesarean section, but commonly staples or dissolvable suture is used. Recently plastic surgeons have found that non-dissolvable suture may have a better cosmetic outcome than staples. The investigators hope to learn if there is a difference in pain both at suture/staple removal and 6 weeks postoperatively between Prolene suture, Absorbable suture (monocryl or vicryl) or staples. The investigators also plan to look for differences in wound complications and patient satisfaction, as well as operating and removal times. This knowledge will be important in helping practitioners choose the closure technique at cesarean delivery.

DETAILED DESCRIPTION:
Patients who meet inclusion criteria will be approached upon admission to Labor and Delivery. A study staff member will describe the study and offer participation. If a patient agrees to participate, she will sign research protocol and HIPAA consent forms and receive a copy of these forms. The patient's chart will be flagged, indicating that she is a study participant. The patient's prenatal care and labor and delivery will be managed by her physician per standard of care at the physician's discretion, including routine surgical preparation and procedures.

When a participating patient is scheduled for a cesarean section, she will be randomized to Arm 1 (Staples) or Arm 2 (Prolene) or Arm 3 (Monocryl or Vicryl absorbable suture). She will be treated as per standard of care and her cesarean section performed per physician discretion. After the closure of the fascial layer, the surgeons will follow the same protocol for each study participant, including wound irrigation with warm sterile saline and reapproximation of the subcutaneous layer if greater than 2.0 cm in depth (per standard of care). The patient in Arm 1 will have skin closure with staples. The patient in Arm 2 will have skin closure with 2-0 Prolene in a subcuticular fashion. The patient in Arm 3 will have skin closure with monocryl or vicryl in the standard fashion. Patients in Arms 1 and 2 will have their closure material removed at the physician's discretion per the standard of care at post-operative day 3 or 4.

Pain level will be assessed on the first and third or fourth day after surgery and again at six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing primary or repeat cesarean section
* Maternal age greater than or equal to 18 years of age
* Gestational age greater than or equal to 34 weeks
* Elective and non-elective cesarean section

Exclusion Criteria:

* Type 1 or Type 2 diabetes
* BMI greater than 35
* Pre-operative diagnosis of chorioamnionitis
* History of drug or alcohol abuse
* Contraindication to NSAIDs
* Chronic pain diagnosis
* Narcotic use prior to pregnancy
* Maternal age less than 18 years of age
* General anesthesia
* Chorioamnionitis, clinical suspicion of chorioamnionitis, or risk factors for chorioamnionitis (membrane rupture greater than 18 hours, GBS positive status)
* Vertical skin incision

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2013-05-04 (Actual); Study Completion 2013-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natali Aziz, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Childrens Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment into the first two arms (Staples and Prolene non-absorbable sutures) occurred through May 2013. The study protocol was modified in July 2014 and the third arm of the study, absorbable sutures, was added, however, no recruitment occurred after this modification.
Period: Overall Study
Arm/Group | Staples | Prolene Non-absorbable Sutures | Absorbable Sutures
Started | 7 | 8 | 0
Completed | 7 | 8 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No enrollment occurred after adding the "absorbable sutures" study arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Staples | Prolene Non-absorbable Sutures | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33.0 [24.5 to 38.5] | 33.5 [31.5 to 34.5] | 33.3 [28 to 36.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 2 | 2 | 4
  Non-Hispanic Black | 0 | 0 | 0
  Hispanic | 2 | 4 | 6
  Asian | 3 | 2 | 5
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain on a Scale During the Post-operative Hospitalization Period
Description: Pain level on a Mosby visual analog pain scale of 1 (no pain) to 10 (worst pain)
Time Frame: Post-operative day 3 or 4.
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 3 | 5
units on a scale | 2.0 [1.5 to 3.4] | 2.0 [2.0 to 2.0]
Statistical Analysis 1: Comparison: Staples vs Prolene Non-absorbable Sutures; Test type: Superiority; p = 0.60, t-test, 2 sided

2. Secondary Outcome: Level of Pain on a Scale at 6 Weeks Postpartum
Description: Pain level on a scale (Mosby visual analog pain scale) of 1 (no pain) to 10 (worst pain).
Time Frame: Post-operative week 6
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 1 | 3
units on a scale | 3 [3 to 3] | 1 [1 to 1]

3. Secondary Outcome: Count of Participants With Wound Complications
Description: Wound complications include conditions like infection, seroma/hematoma and dehiscence
Time Frame: Post-operative week 6
Population: Only patients with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 1 | 3
Participants | 0 | 0

4. Secondary Outcome: Level of Patient Satisfaction to the Wound Appearance
Description: Level of patient satisfaction measured on a scale of 1 (very unsatisfied) to 10 (very satisfied)
Time Frame: Post-operative day 3 or 4
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 0 | 3
units on a scale |  | 9 [8.5 to 9.0]

5. Secondary Outcome: Level of Patient Satisfaction to the Wound Appearance at 6 Weeks Postpartum
Description: Level of patient satisfaction measured on a scale of 1 (very unsatisfied) to 10 (very satisfied)
Time Frame: Post-operative week 6
Population: There were no patients that had data available for analysis for "staples" and "prolene non-absorbable sutures" study arms.
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time From Skin Incision to the Skin Closure
Description: Measured in minutes
Time Frame: Day of cesarean delivery (up to 8 hours)
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 7 | 8
minutes | 55.0 [46.0 to 61.0] | 56.5 [54.0 to 62.25]

7. Secondary Outcome: Time Needed for the Suture Removal
Description: Measured in seconds
Time Frame: Post-operative day 3 or 4
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 2 | 4
seconds | 79.0 [73.5 to 84.5] | 1.5 [1.0 to 1.75]

8. Secondary Outcome: Level of Patient's Satisfaction to the Cosmesis of the Wound
Description: Measured on a scale of 0 (very unsatisfied to the cosmesis) to 10 (very satisfied to the cosmesis)
Time Frame: Post-operative week 6
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 5 | 3
units on a scale | 9.0 [8.0 to 10.0] | 5.0 [5.0 to 7.5]

9. Secondary Outcome: Level of Patient's Overall Patient Satisfaction to the Type of Closure
Description: Level of patient satisfaction measured on a scale of 1 (very unsatisfied) to 10 (very satisfied)
Time Frame: Post-operative day 1
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 2 | 2
units on a scale | 8.0 [7.5 to 8.5] | 7.5 [6.25 to 8.75]

10. Secondary Outcome: Level of Patient's Overall Patient Satisfaction to the Type of Closure
Description: Level of patient satisfaction measured on a scale of 1 (very unsatisfied) to 10 (very satisfied)
Time Frame: Post-operative day 3 or 4
Population: Only patients with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 0 | 3
units on a scale |  | 8.7 [8.5 to 9.0]

11. Secondary Outcome: Level of Patient's Overall Patient Satisfaction to the Type of Closure
Description: Level of patient satisfaction measured on a scale of 1 (very unsatisfied) to 10 (very satisfied)
Time Frame: Post-operative week 6
Population: No patients had data available for the analysis.
Arm/Group | Staples | Prolene Non-absorbable Sutures
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 weeks after cesarean delivery.
Arm/Group | Staples | Prolene Non-absorbable Sutures
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes